CLINICAL TRIAL: NCT02484352
Title: Optimal Dose of Intravenous Oxycodone for Attenuation of Hemodynamic
Brief Title: Optimal Dose of Intravenous Oxycodone for Endotracheal Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yong-Hee Park (Other)
Collaborators: Chung-Ang University (Other)
Responsible Party: Sponsor-Investigator, Yong-Hee Park, Assistant professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Organization: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C2014115(1311)
Record Dates: First submitted 2015-06-19; First posted 2015-06-29 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Intubation Complication; Blood Pressure
Keywords: dosage of oxycodone during intubation
MeSH Terms: interventions — Sodium Chloride; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0 mg/kg of oxycodone (Other): Intervention: patients receive 10 ml of normal saline without oxycodone through intravenous route before intubation.
  Interventions: Drug: saline
- 0.05 mg/kg of oxycodone (Other): Intervention: patients receive 10 ml of fluid with 0.05 mg/kg of oxycodone in normal saline through intravenous route before intubation.
  Interventions: Drug: 0.05 mg/kg of oxycodone
- 0.1 mg/kg of oxycodone (Other): Intervention: patients receive 10 ml of fluid with 0.1 mg/kg of oxycodone in normal saline through intravenous route before intubation.
  Interventions: Drug: 0.1 mg/kg of oxycodone
- 0.15 mg/kg of oxycodone (Other): Intervention: patients receive 10 ml of fluid with 0.15 mg/kg of oxycodone in normal saline through intravenous route before intubation.
  Interventions: Drug: 0.15 mg/kg of oxycodone
- 0.2 mg/kg of oxycodone (Other): Intervention: patients receive 10 ml of fluid with 0.2 mg/kg of oxycodone in normal saline through intravenous route before intubation.
  Interventions: Drug: 0.2 mg/kg of oxycodone

INTERVENTIONS:
Drug: saline — different dosage of IV oxycodone was given before intubation
  Arms: 0 mg/kg of oxycodone
Drug: 0.05 mg/kg of oxycodone — different dosage of IV oxycodone was given before intubation
  Other Names: OxyNorm
  Arms: 0.05 mg/kg of oxycodone
Drug: 0.1 mg/kg of oxycodone — different dosage of IV oxycodone was given before intubation
  Other Names: OxyNorm
  Arms: 0.1 mg/kg of oxycodone
Drug: 0.15 mg/kg of oxycodone — different dosage of IV oxycodone was given before intubation
  Other Names: OxyNorm
  Arms: 0.15 mg/kg of oxycodone
Drug: 0.2 mg/kg of oxycodone — different dosage of IV oxycodone was given before intubation
  Other Names: OxyNorm
  Arms: 0.2 mg/kg of oxycodone

SUMMARY:
Intravenous form of oxycodone is recently used for the adjunct of anesthetic agents to avoid adverse effects of the stimulation of endotracheal intubation. The potency ratio of oxycodone to fentanyl is not absolutely defined. The aim of this study was to assess the optimal dose of intravenous oxycodone for attenuation of hemodynamic responses to laryngoscopy and endotracheal intubation.

A prospective, randomized, double-blind study was conducted. Ninety one patients were randomly divided into 5 group based on the dose of oxycodone; 0, 0.05, 0.1, 0.15, 0.2 mg/kg. After giving each assigned dose of intravenous oxycodone, anesthesia was induced with thiopental and rocuronium. Heart rate (HR) and blood pressure (BP) was collected at baseline, before intubation, 1, 2, 3 minutes after intubation. The change of BP was calculated by (highest BP after intubation - baseline BP)/baseline BP.

DETAILED DESCRIPTION:
Endotracheal intubation is almost always associated with increase of catecholamine and arterial blood pressure. To prevent the responses to laryngoscopy and tracheal intubation, adjuvant use of opioid to sedative drugs during anesthetic induction phase are common. Intravenous form of oxycodone is recently used for the adjunct of anesthetic agents to avoid adverse effects of the stimulation of endotracheal intubation. However, The potency ratio of oxycodone to fentanyl is not absolutely defined. Therefore, the investigators aimed to assess the optimal dose of intravenous oxycodone for attenuation of hemodynamic responses to laryngoscopy and endotracheal intubation.

The patients were randomly divided into five different groups based on the dose of oxycodone; 0. 0.05, 0.1, 0.15, 0.2 mg/kg. The drug was prepared by a person who is not participating the anesthetic management and surgery of the patient. In five groups, the drug was mixed with normal saline which makes the total drug volume to be 10 ml. After monitoring was started including ECG, noninvasive blood pressure, and pulse oximetry, the anesthesiologist who has no information about the drug give the drug when starting induction of anesthesia. Thiopental 4-5 mg/kg and rocuronium 0.6-0.9 mg/kg was given subsequently. Manual ventilation was done with sevoflurane 3-5 volume% for 2-3 minutes and tracheal intubation was done. Maintenance of anesthesia was done with 50% O2 with nitrous oxide and sevoflurane. Mechanical ventilation was done with tidal volume 10 ml/kg and respiratory rate 12 /min. The baseline hemodynamic data including heart rate and blood pressure was recorded and those before intubation, 1,2,3 minutes after intubation were obtained. The discrepancies between the highest and baseline, the lowest blood pressure and heart rate and baseline were used to make out the proportion of hemodynamic changes. This proportion of the hemodynamic changes were compared in five groups. In addition, the use of vasopressor was also recorded and the frequency and the cumulative dose was compared among the groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 1

Exclusion Criteria:

* ASA class over 2
* expected difficult intubation
* intubation time over 30 seconds
* intubation trial was more than once

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2017-02-12 (Actual)

PRIMARY OUTCOMES:
blood pressure changes before and after endotracheal intubation | from entrance to operating room to intubation time; up to 30 minutes
  highest blood pressure and baseline blood pressure

SECONDARY OUTCOMES:
total dose of vasopressor; dose x frequency | during the induction phase of anesthesia before surgical incision up to 30 minutes
heart rate changes before and after endotracheal intubation | from entrance to operating room to intubation time; up to 30 minutes
  highest heart rate and baseline heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Young-Cheol Woo, Ph.D., Study Director — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine : Chung-Aung University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sawano Y, Miyazaki M, Shimada H, Kadoi Y. Optimal fentanyl dosage for attenuating systemic hemodynamic changes, hormone release and cardiac output changes during the induction of anesthesia in patients with and without hypertension: a prospective, randomized, double-blinded study. J Anesth. 2013 Aug;27(4):505-11. doi: 10.1007/s00540-012-1552-x. Epub 2013 Jan 12. PMID 23314694
- [Background] Russell WJ, Morris RG, Frewin DB, Drew SE. Changes in plasma catecholamine concentrations during endotracheal intubation. Br J Anaesth. 1981 Aug;53(8):837-9. doi: 10.1093/bja/53.8.837. PMID 7272146